CLINICAL TRIAL: NCT02047682
Title: Implementation of Physical Exercise at the Workplace (IRMA10) - Occupational Load
Acronym: IRMA10
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Southampton (Other)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, PhD, National Research Centre for the Working Environment, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRMA10
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Musculoskeletal Disorders; Stress
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Models, Biopsychosocial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biopsychosocial (Experimental): Biopsychosocial intervention with Individually tailored physical exercises and stress management
  Interventions: Behavioral: Biopsychosocial
- Reference (Active Comparator): Reference group receiving "usual care" in terms of standard workplace ergonomics and physical exercises
  Interventions: Behavioral: Reference

INTERVENTIONS:
Behavioral: Biopsychosocial
  Arms: Biopsychosocial
Behavioral: Reference
  Arms: Reference

SUMMARY:
Static postures, repetitive work tasks, and work stress increase the risk for musculoskeletal disorders and sickness absence. Objective measurements of occupational loadings - EMG for muscular activity, EEG for cognitive activity, ECG for cardiovascular activity and heart rate variability, actigraphy for bodily movements - may provide useful early indicators of muscular, cognitive and cardiovascular overload.

The aim of this study is to investigate the effect of an individually tailored bio-psycho-social intervention strategy versus "usual care" ergonomics and standard physical exercises (reference group) on these risk factors in lab technicians with a history of work-related musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory technician
* Pain intensity >= 3 (scale of 0-10)
* Pain duration >= 3 months
* Pain frequency >= 3 days per week

Exclusion Criteria:

* life threatening disease
* pregnancy

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
EMG gaps | change from baseline to week 10
  Electromyography (EMG) is measured in the neck and shoulder muscles throughout a normal workday before and after the intervention. EMG gaps is defined as periods with muscular inactivity. Actigraphs are used to measure bodily movements, and only period with sitting or standing work are included in the analysis (i.e. walking activities are excluded from the analyses)

SECONDARY OUTCOMES:
EEG | change from baseline to week 10
  Electroencephalography is measured throughout a normal workday before and after the intervention. Actigraphs are used to measure bodily movements, and only period with sitting or standing work are included in the analysis (i.e. walking activities are excluded from the analyses)
HRV | change from baseline til 10 week followup
  Heart Rate Variability (HRV) is measured with Actiheart throughout the working day before and after the intervention. Actigraphs are used to measure bodily movements, and only period with sitting or standing work are included in the analysis (i.e. walking activities are excluded from the analyses)

CONTACTS AND LOCATIONS:
Overall Officials: Lars L Andersen, PhD, Principal Investigator — National Research Centre for the Working Environment, Denmark
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark